CLINICAL TRIAL: NCT02684591
Title: Aramchol Versus Placebo in the Treatment of HIV-associated Nonalcoholic Fatty Liver Disease and Lipodystrophy: A Randomized, Double-blinded, Allocation-concealed, Placebo-controlled Clinical Trial
Brief Title: Aramchol for HIV-associated Nonalcoholic Fatty Liver Disease and Lipodystrophy
Acronym: ARRIVE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Rohit Loomba, Professor of Medicine, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ARRIVE
Record Dates: First submitted 2016-01-15; First posted 2016-02-18 (Estimated); Results first posted 2019-08-21 (Actual); Last update posted 2020-07-17 (Actual); Status verified 2020-07

CONDITIONS: Nonalcoholic Fatty Liver Disease; HIV
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease | interventions — aramchol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Aramchol 600 mg orally daily (Experimental): Total 600 mg Aramchol (200 mg/tablet and 400 mg/tablet) per day once a day orally for 12 weeks.
  Intervention: Aramchol
  Interventions: Drug: Aramchol
- Placebo (Placebo Comparator): Placebo in the form of a tablet; Two bottles will be given to patient and they will take two pills, once a day orally for 12 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Aramchol — Aramchol, a conjugate of Cholic acid and Arachidic acid, is a first in class member of a novel family of synthetic Fatty-Acid / Bile-Acid Conjugates (FABACs). FABACs are composed of endogenic compounds, orally administrated with potentially good safety and tolerability parameters
  Other Names: arachidyl amido cholanoic acid
  Arms: Aramchol 600 mg orally daily
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
A subset of patients with NAFLD that have not been extensively studied are those infected with human immunodeficiency virus (HIV). Currently, there is no FDA approved treatment for NAFLD or NASH. Additionally, there have been no significant clinical trials for HIV patients with NAFLD and there are no approved treatment options. We plan to conduct a randomized, double-blinded, placebo-controlled clinical trial to examine the efficacy of 600 mg of Aramchol daily (including 200 mg tablet and 400 mg tablet) versus identical placebo given over 12 weeks to improve HIV-associated hepatic steatosis as measured by a validated and accurate magnetic resonance imaging (MRI)-based technique.

DETAILED DESCRIPTION:
We plan to conduct a randomized, double-blinded, placebo-controlled clinical trial to examine the efficacy of Aramchol at 600 mg/day orally versus identical placebo given over 12 weeks to improve HIV-associated hepatic steatosis as measured by a validated and accurate magnetic resonance imaging (MRI)-based technique. In this study, we propose to randomize up to 50 patients with HIV-associated NAFLD to either Aramchol or placebo for 12 weeks. We plan to enroll a total of 55 patients, expecting some drop outs prior to randomization. After an initial evaluation for insulin sensitivity, liver fat measurement by MRI, and total body fat content by DEXA, patients will be randomized to receive either Aramchol 600 mg/day or placebo orally for 12 weeks. Patients will be monitored at regular intervals for symptoms of liver disease, side effects of medication, and serum biochemical and metabolic indices. Patients will also be assessed for continued HIV viral load suppression and continued tolerance of antiretroviral therapy. At the end of 12 weeks, patients will have a repeat medical evaluation, liver fat measurement, and total body fat content measurement. Pre and post treatment liver fat by MRI, ALT/AST, HbA1c, CRP, insulin sensitivity, and DEXA for whole body fat will be compared. The primary end point of successful therapy will be improvement in liver fat by MRI. Secondary end points will be improvement in total body fat, insulin sensitivity and liver biochemistry.

ELIGIBILITY:
Inclusion Criteria:

1. Age at entry at least 18 years.
2. And at least one of the following risk factor for more severe liver disease: Hypertriglyceridemia based upon ATP-III guidelines, Increased LDL cholesterol or increased total cholesterol based upon ATP-III guidelines, Decreased HDL cholesterol based upon ATP-III guidelines, Serum alanine (ALT) or aspartate (AST) aminotransferase activities that are above the upper limits of normal. 19 or more in women and 30 or more in men, Overweight as defined as BMI: 25 < 30 kg/m2, Obesity as defined BMI ≥ 30 kg/m2, Hyperuricemia based upon ATP-III guidelines, Prediabetes or Diabetes by American Diabetes Association Criteria
3. Lipodystrophy will be confirmed on both clinical and radiologic assessment and defined as: Clinical history and/or exam by the study physician with signs of either facial,temporal, upper or lower extremity lipo-atrophy, Documented abdominal fat accumulation with presence of hepatic steatosis on MRI
4. An MRI-determined fat fraction classification threshold (≥5%) will be used to confirm subjects. MR examinations will include four research sequences (three imaging sequences and one single-voxel spectroscopy sequence) that have been developed and refined by Dr. Sirlin, allowing for the measurement of liver fat fraction and newer candidate MR biomarkers for future NAFLD studies. MR examinations will last 20-30 minutes and will be performed without contrast agents. Subjects will be scanned at 1.5T. To assess sequence repeatability, two sequences per subject, block randomized, will be run three times. For MR elastography, MR imaging will be done which will include placing a vibrating paddle over the abdomen while images are obtained. A comprehensive screening questionnaire will be utilized prior to subjects having an MRI. Experienced research MR technologists will perform MR examinations under the supervision of Dr. Sirlin.
5. History of HIV documented by a previously positive HIV Elisa or PCR.
6. Stable antiretroviral (ART) regimen for at least 12 weeks prior to study inclusion.
7. Written informed consent.

Exclusion Criteria:

1. Evidence of another form of liver disease: Hepatitis B as defined as presence of hepatitis B surface antigen (HBsAg), Hepatitis C as defined by presence of hepatitis C virus (HCV) RNA in serum, Autoimmune hepatitis as defined by anti-nuclear antibody (ANA) of 1:160 or greater and liver histology consistent with autoimmune hepatitis or previous response to immunosuppressive therapy, Autoimmune cholestatic liver disorders as defined by elevation of alkaline phosphatase and anti-mitochondrial antibody of greater than 1:80 or liver histology consistent with rimary biliary cirrhosis or elevation of alkaline phosphatase and liver histology consistent with sclerosing cholangitis, Wilsons disease as defined by ceruloplasmin below the limits of normal and liver histology consistent with Wilsons disease Alpha-1-antitrypsin deficiency as defined by alpha-1-antitrypsin level less than normal and liver histology consistent with alpha-1-antitrypsin deficiency hemochromatosis as defined by presence of 3+ or 4+ stainable iron on liver biopsy and homozygosity for C282Y or compound heterozygosity for C282Y/H63D, Drug-induced liver disease as defined on the basis of typical exposure and history,Bile duct obstruction as shown by imaging studies.
2. Evidence of liver cirrhosis based upon clinical assessment, imaging or any of the following lab abnormalities: INR >1.4, albumin <3.2 g/dL, platelet count <90 x 103/microliter
3. History of excess alcohol ingestion, averaging more than 30 gm/day (3 drinks per day) in the previous 10 years, or history of alcohol intake averaging greater than 10 gm/day (1 drink per day or 7 drinks per week) in the previous one year.
4. Contraindications to MRI: The subject has any contraindication to MR imaging, such as patients with pacemakers, metallic cardiac valves, magnetic material such as surgical clips, implanted electronic infusion pumps or other conditions that would preclude proximity to a strong magnetic field, the subject has a history of extreme claustrophobia, The subject cannot fit inside the MR scanner cavity, decompensated liver disease, Child-Pugh score greater than or equal to 7 points

6. History of gastrointestinal bypass surgery or ingestion of drugs known to produce hepatic steatosis including corticosteroids, high-dose estrogens, methotrexate, tetracycline or amiodarone in the previous 6 months. 7. Recent use (within the last 90 days) of medications to treat hepatic steatosis such as pioglitazone (or medications in the same class) or vitamin E. 8. Use of Aramchol or agents in the same class. 9. Recent use (within the last 90 days) of insulin as an outpatient for management of diabetes.

10. HbA1c > 9 or uncontrolled diabetes. 11. Significant systemic or major illnesses other than liver disease, including congestive heart failure, coronary artery disease, cerebrovascular disease, pulmonary disease with hypoxia, renal failure, organ transplantation, serious psychiatric disease, malignancy that, in the opinion of the investigator would preclude treatment with Aramchol and adequate follow up.

12. Active substance abuse, such as alcohol, inhaled or injection drugs within the previous one year. 13. Pregnancy or inability to practice adequate contraception in women of childbearing potential.

14. Evidence of hepatocellular carcinoma: alpha-fetoprotein levels greater than 200 ng/ml and/or liver mass on imaging study that is suggestive of liver cancer.

15. HIV specific exclusions: CD4 count of less than 200 cells/μL, Detectable viral load,Changes to ART regimen in the preceding 12 weeks,Lack of alternative ART regimens should the patient experience virologic breakthrough,History of opportunistic infection in the preceding 12 months

16. Symptoms of uncontrolled gastrointestinal disorders involving motility, gastric acid or gastric emptying malabsorption ,Disorders including but not limited to peptic ulcer disease, gastroesophageal reflux, dyspepsia, gastroparesis, chronic diarrhea, chromic constipation, gall bladder disease,pancreatitis, lactose intolerance and celiac disease.Patients who have used anticholinergic or other drugs known to affect gastrointestinal motility within 7 days prior to dosing and throughout the study will also be excluded

17. Patients with hypersensitivity to Aramchol or to any of the excipients in the tablets or with hypersensitivity to cholic acid or bile acid sequestrants

18. Any other condition, which, in the opinion of the investigators would impede competence or compliance or possibility hinder completion of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2016-01; Primary Completion 2018-02 (Actual); Study Completion 2018-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rohit Loomba, M.D., Principal Investigator — University of California, San Diego
Locations (1):
- University of California, San Diego, San Diego, California, United States

REFERENCES:
- [Derived] Ajmera VH, Cachay E, Ramers C, Vodkin I, Bassirian S, Singh S, Mangla N, Bettencourt R, Aldous JL, Park D, Lee D, Blanchard J, Mamidipalli A, Boehringer A, Aslam S, Leinhard OD, Richards L, Sirlin C, Loomba R. MRI Assessment of Treatment Response in HIV-associated NAFLD: A Randomized Trial of a Stearoyl-Coenzyme-A-Desaturase-1 Inhibitor (ARRIVE Trial). Hepatology. 2019 Nov;70(5):1531-1545. doi: 10.1002/hep.30674. Epub 2019 Jun 18. PMID 31013363

RESULTS

PARTICIPANT FLOW:
Groups:
- Aramchol 600 mg Orally Daily: Total 600 mg Aramchol (200 mg/tablet and 400 mg/tablet) per day once a day orally for 12 weeks.
  Intervention: Aramchol
  Aramchol: Aramchol, a conjugate of Cholic acid and Arachidic acid, is a first in class member of a novel family of synthetic Fatty-Acid / Bile-Acid Conjugates (FABACs). FABACs are composed of endogenic compounds, orally administrated with potentially good safety and tolerability parameters
Period: Overall Study
Arm/Group | Aramchol 600 mg Orally Daily | Placebo
Started | 25 | 25
Completed | 24 | 22
Not Completed | 1 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Aramchol 600 mg Orally Daily | Placebo | Total
Number analyzed (Participants) | 25 | 25 | 50
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.6 (11.4) | 49.7 (9.0) | 48.2 (10.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 1 | 4
  Male | 22 | 24 | 46
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 11 | 6 | 17
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 14 | 19 | 33
MRI PDFF - Magnetic resonance imaging proton density fat fraction [Median (Full Range); unit: percentage of fat] | 16.2 [5.4 to 31.6] | 12.1 [5.4 to 40.1] | 12.8 [5.4 to 40.1]

OUTCOME MEASURES:

1. Primary Outcome: Efficacy of Aramchol 600 mg vs. Placebo in Improving Hepatic Steatosis Assessed by Magnetic Resonance Imaging in Patients With HIV-associated NAFLD
Description: To examine the efficacy of aramchol at 600 mg orally daily versus placebo in improving hepatic steatosis assessed by magnetic resonance imaging in patients with HIV-associated NAFLD
Time Frame: 12 weeks
Measure: Median (Full Range); unit: percentage of fat
Arm/Group | Aramchol 600 mg Orally Daily | Placebo
Number analyzed (Participants) | 24 | 22
percentage of fat | 13.7 [1.5 to 26.3] | 11.1 [2.7 to 24.3]

2. Secondary Outcome: Serum Alanine Aminotransferase (ALT)
Description: To examine the efficacy of two doses of aramchol: 200 mg/tablet and 400 mg/tablet / day orally daily versus placebo in improving serum alanine aminotransferase (ALT) levels in patients with HIV-associated NAFLD
Time Frame: 12 Weeks
Measure: Median (Full Range); unit: IU/L
Arm/Group | Aramchol 600 mg Orally Daily | Placebo
Number analyzed (Participants) | 24 | 22
IU/L | 51 [12 to 100] | 35 [14 to 83]

ADVERSE EVENTS:
Time Frame: 12 Weeks
Arm/Group | Aramchol 600 mg Orally Daily | Placebo
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/25
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/25
Other Adverse Events (participants affected / at risk) | 4/25 | 3/25
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Aramchol 600 mg Orally Daily (N=25) | Placebo (N=25)
Acid Reflux (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal Pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Cellulitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2011-05-11): https://cdn.clinicaltrials.gov/large-docs/91/NCT02684591/Prot_SAP_000.pdf